CLINICAL TRIAL: NCT01594983
Title: A Multicenter, Randomized, Active Comparator, Placebo Controlled, Double-blind Pilot Study to Assess the Efficacy and Safety of LCQ908 Alone and in Combination With Fenofibrate or Lovaza® in Patients With Severe Hypertriglyceridemia
Brief Title: A Pilot Study to Assess the Efficacy and Safety of LCQ908 Alone and in Combination With Fenofibrate or Lovaza® in Patients With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCQ908C2201; 2012-000872-40 (EudraCT Number)
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2015-10

CONDITIONS: Non Familial Chylocmicronemia Syndrome (Non-FCS)
Keywords: hypertriglyceridemia; Non familial Chylocmicronemia Syndrome (non-FCS)
MeSH Terms: conditions — Hypertriglyceridemia | interventions — pradigastat; Fenofibrate; Fish Oils; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- LCQ908 1 (Experimental): LCQ908 (Diacylglycerol acyltransferase inhibitor)once daily for 12 weeks
  Interventions: Drug: LCQ908; Drug: Placebo of LCQ908; Drug: Placebo of fenofibrate; Drug: Placebo of fish oil
- LCQ908 2 (Experimental): LCQ908 once daily for 12 weeks
  Interventions: Drug: LCQ908; Drug: Placebo of LCQ908; Drug: Placebo of fenofibrate; Drug: Placebo of fish oil
- LCQ908 3 (Experimental): LCQ908 once daily for 12 weeks
  Interventions: Drug: LCQ908; Drug: Placebo of LCQ908; Drug: Placebo of fenofibrate; Drug: Placebo of fish oil
- Fenofibrate (Active Comparator): Intervention Type: Drug Intervention Name: Fenofibrate
  Interventions: Drug: LCQ908; Drug: Fenofibrate; Drug: Placebo of LCQ908; Drug: Placebo of fish oil
- Fish Oil (Active Comparator): Fish oil once daily for 12 weeks
  Interventions: Drug: LCQ908; Drug: Fish Oil; Drug: Placebo of LCQ908; Drug: Placebo of fenofibrate
- Arm Label: Placebo (Placebo Comparator): Intervention Type: other Intervention Name: other
  Interventions: Drug: Placebo of LCQ908; Drug: Placebo of fenofibrate; Drug: Placebo of fish oil

INTERVENTIONS:
Drug: LCQ908
  Arms: Fenofibrate; Fish Oil; LCQ908 1; LCQ908 2; LCQ908 3
Drug: Fenofibrate — Fenofibrate once daily 12 weeks
  Arms: Fenofibrate
Drug: Fish Oil — Fish Oil once daily for 12 weeks
  Other Names: Lovaza®
  Arms: Fish Oil
Drug: Placebo of LCQ908 — Matching placebo of LCQ908
Drug: Placebo of fenofibrate — Matching placebo of fenofibrate
  Arms: Arm Label: Placebo; Fish Oil; LCQ908 1; LCQ908 2; LCQ908 3
Drug: Placebo of fish oil — Matching placebo of fish oil capsule
  Arms: Arm Label: Placebo; Fenofibrate; LCQ908 1; LCQ908 2; LCQ908 3

SUMMARY:
This study is to determine a dose response signal for LCQ908 monotherapy and to assess the efficacy and safety of adding LCQ908 to Lovaza or fenofibrate.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages >18 years of age, inclusive.
* History of plasma TG concentration ≥890 mg/dl (10 mmol/L) or history of lactescent plasma in the fasting state.
* Fasting TG ≥ 750 mg/dL (8.5 mmol/L) at day -7 or repeat of day -7 one week later for those failing to qualify initially and thought likely to qualify on repeat examination prior to randomization.

Exclusion Criteria:

* Treatment with Omega-3 fatty acids or niacin or fibrates within 8 weeks of screening.
* Patients with confirmed Familial Chylomicronemia Syndrome (FCS) with hyperlipoproteinemia (HLP) Type-I diagnosis or known to be homozygotes or compound heterozygotes for mutations in HLP Type I-causing genes (such as LPL, apoCII, CPIHBP1, or LMF1) prior to screening.
* Pancreatitis within 3 months prior to screening.
* Uncontrolled type 2 diabetes (T2DM) (as defined by an HbA1c value of ≥8.0% at screening)
* BMI > 40 or history of bariatric surgery.
* Nephrotic syndrome, Type 1 diabetes, HIV, HCV or HBV positive.
* Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73m2

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in triglycerides (TG) relative to placebo at 6 weeks | Baseline, 6 weeks
  The dose response signal of 3 dose regiments of LCQ908 in patients at risk for non-FCS chylomicronemia as was measured by change from baseline in triglycerides (TG) relative to placebo at 6 weeks.

SECONDARY OUTCOMES:
Change from baseline in triglycerides after adding LCQ908 to background therapy of fenofibrate or Fish Oil at 12 weeks | Baseline, 12 weeks
Changes from baseline in triglycerides after treatment with LCQ908 monotherapy relative to fenofibrate or fish oil at 6 weeks | Baseline, 6 weeks
Change from baseline in triglycerides after treatment with LCQ908 monotherapy relative to placebo at 12 weeks | Baseline, 12 weeks
Number of patients in LCQ908 monotherapy with adverse events , serious adverse events and death | 12 weeks
changefrom baseline in lipids and lipoprotein profiles | Baseline, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (26):
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Orange City, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Oxon Hill, Maryland
  - Novartis Investigative Site, Butte, Montana
  - Novartis Investigative Site, Cary, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Lyndhurst, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Lansdale, Pennsylvania
  - Novartis Investigative Site, Bristol, Tennessee
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, Corpus Christi, Texas
  - Novartis Investigative Site, Houston, Texas
- Canada (2):
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- See also: Results for CLCQ908C2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12104